CLINICAL TRIAL: NCT07405281
Title: A Multicenter, Prospective Clinical Randomized Controlled Study of the Efficacy of Hyperbaric Oxygen on Acute Ankle Sprain
Brief Title: the Efficacy of Hyperbaric Oxygen on Acute Ankle Sprain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2025-1461
Record Dates: First submitted 2026-01-20; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Ankle Sprain
Keywords: acute ankle sprain; hyperbaric oxygen
MeSH Terms: conditions — Ankle Injuries | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hyperbaric oxygen group (Experimental): The treatment is administered at an atmospheric pressure of 2 ATA, with 100% oxygen inhalation.
  Interventions: Other: hyperbaric oxygen therapy
- non hyperbaric oxygen group (Sham Comparator): The treatment is administered at an atmospheric pressure of 1.4 ATA with an inhaled oxygen fraction of 21%
  Interventions: Other: non Hyperbaric Oxygen Therapy

INTERVENTIONS:
Other: hyperbaric oxygen therapy — The treatment is administered at an atmospheric pressure of 2 ATA, with 100% oxygen inhalation. Oxygen inhalation time: 40 minutes (inhaling oxygen for 20 minutes, resting for 5 minutes, inhaling oxygen for 20 minutes, decompression), once daily, for 14 consecutive days. (Commenced immediately after randomisation)
  Arms: hyperbaric oxygen group
Other: non Hyperbaric Oxygen Therapy — The treatment is administered at an atmospheric pressure of 1.4 ATA with an inhaled oxygen fraction of 21%, oxygen inhalation time: 40 minutes (20 minutes of oxygen inhalation, 5 minutes rest, 20 minutes of oxygen inhalation, decompression), once daily, for 14 consecutive days. (Commences immediately after randomisation)
  Arms: non hyperbaric oxygen group

SUMMARY:
Investigators recruited 208 patients with acute ankle sprain who were from the Rehabilitation Department of the Second Affiliated Hospital of Zhejiang University, School of Medicine from January 2026 to November 2028. Perform the improvement in AOFAS scores and Baird-Jackson ankle scores study and Rehabilitation assessments followed up after 3 years.

DETAILED DESCRIPTION:
In baseline, 208 patients with i acute ankle sprain were recruited from the Rehabilitation Department of the Second Affiliated Hospital of Zhejiang University School of Medicine from January 2026 to December 2028, and were followed up after 3 years.

Perform the improvement in AOFAS scores and Baird-Jackson ankle scores study and Rehabilitation assessments followed up after 3 years. The Hyperbaric oxygen group treatment was administered at an atmospheric pressure of 2 ATA, with 100% oxygen inhalation. Oxygen was inhaled for 40 minutes (20 minutes of oxygen inhalation, 5-minute rest, 20 minutes of oxygen inhalation, decompression), once daily for 14 consecutive days. The control group treatment at an atmospheric pressure of 1.4 ATA, inhaling 21% oxygen by volume. Oxygen inhalation schedule: 40 minutes (inhale oxygen for 20 minutes, rest for 5 minutes, inhale oxygen for 20 minutes, decompression), once a day for 14 consecutive days.

Two person analyzed the above data, and record abnormal results.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral ankle sprain;
* Swelling, bruising, and pain at the site of the sprain;
* Injury occurring within 72 hours;
* MRI examination clearly shows ligament damage.

Exclusion Criteria:

* X-ray shows ankle fracture;
* Ankle has skin lesions or skin diseases;
* History of lower limb and pelvic surgery;
* Obvious neurological or psychiatric disorders that may interfere with assessment;
* Severe ligament injuries or joint instability requiring surgical treatment;
* Previous ankle injuries, persistent pain or functional limitations;
* Pneumothorax, severe emphysema, active bleeding, or other diseases with contraindications for hyperbaric oxygen therapy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 208 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2029-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
AOFAS score | 3 years
  Improvement of American Orthopaedic Foot & Ankle Society Score （AOFAS scores）in acute ankle sprains with early HBO treatment. Usually scored from 0 to 100, higher scores mean a better outcome.
Baird-Jackson ankle score | 3 years
  Improvement of Baird-Jackson Ankle Evaluation Score（Baird-Jackson ankle scores） in acute ankle sprains with early HBO treatment. Usually scored from 0 to 100., higher scores mean a better outcome.

SECONDARY OUTCOMES:
pain scores | 3 years
  The effects of hyperbaric oxygen on improvements in pain scores Visual Analog Scale (VAS) (resting VAS and walking VAS) in patients with acute ankle sprain. Usually scored from 0 to 10. higher scores mean a worth outcome.
ankle swelling | 3 years
  Measure the ankle joint circumference at the level of the medial malleolus tip, in millimeters, on both the affected and healthy sides, and calculate the degree of swelling. The more swollen the joints, the worth the outcome.
high-frequency ultrasound findings | 3 years
  Observe the damage and healing of ligaments and surrounding tissues. The better the continuity of the ligaments and surrounding tissues, the better the outcome.
Ankle MRI | 3 years
  Observe the damage and healing of ligaments and surrounding tissues. The higher the MRI signal, the worse the outcome.
patient's overall evaluation of treatment (PGIC) | 3 years
  The doctor asks the patient about their overall feeling regarding the treatment: 'Has there been any improvement?' Choose one as your answer:
  Number 1 indicates significant improvement; Number 2 indicates slight improvement; Number 3 indicates no change; Number 4 indicates worsening due to the treatment. higher scores mean a worth outcome.
HAMA scale score | 3 years
  the effects of hyperbaric oxygen on change in Hamilton Anxiety Scale（HAMA scale score）in patients with acute ankle sprain. Each item is rated on a five-point scale from 0 to 4. The total score reflects the overall severity of anxiety and can be used to assess treatment effects and changes in the condition.
  Total score ≥29: Possible severe anxiety. Total score ≥21: Definitely significant anxiety. Total score ≥14: Definitely anxiety. Total score ≥7: Possible anxiety. Total score <7: No anxiety symptoms. higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Bing Xiong, Principal Investigator — 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China

IPD SHARING:
Plan to Share IPD: No